CLINICAL TRIAL: NCT05090696
Title: Efficacy and Tolerance Study on the Use of the In-exsufflator in the Hospitalized Elderly
Acronym: INEXPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 ESTENNE (INEXPA); 2021-A00891-40 (Other: 2021-A00891-40)
Record Dates: First submitted 2021-09-16; First posted 2021-10-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Airway Obstruction
Keywords: Airway Obstruction; Mechanical Insufflator Exsufflator; Older Adults
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group only: Participants recruited from patients hospitalized in intensive care units and pulmonary unit of the University Hospital of Clermont-Ferrand, France.
  Interventions: Device: Mechanical In-Exsufflator (MI-E)

INTERVENTIONS:
Device: Mechanical In-Exsufflator (MI-E) — The feasibility will be estimated by quantifying relief and discomfort of four MI-E sessions (2 days x 2 sessions = 4 sessions). Vital signs will be also noted before and after such MI-E session.
  Other Names: Cough Assist

SUMMARY:
The mechanical in-exsufflator (MI-E) is a medical device used to facilitate coughing when the patients' cough is not efficient. Studies have shown positive results in helping airway clearance in children and adults with neuromuscular disorders however there is lack of evidence in older populations. This study's aim is to evaluate the feasibility of the MI-E in older adults. The hypothesis is that the use of MI-E in older adults is feasible.

DETAILED DESCRIPTION:
Background: One of the most frequent reasons for hospital admission of older adults are respiratory disorders. Physiological aging processes decrease respiratory muscle strength and can reduce the efficacity of cough. The mechanical in-exsufflator (MI-E) is a medical device used to help coughing. Studies have shown positive results in helping airway clearance in children and adults with neuromuscular pathologies however there is lack of evidence in older populations. This study's aim is to evaluate the feasibility of the MI-E in older adults. The hypothesis is that the use of MI-E in older adults is feasible.

Methods: Feasibility will be evaluated by outcomes such as the discomfort of each session (use of a numerical scale of discomfort from 0 to 10) and the relief felt before and after each session (use of a modified Borg scale to quantify dyspnea). Two sessions a day of MI-E will be done for a total of four sessions. Furthermore, other outcomes shall be used, before and after each session, such as vital signs (heart and respiratory rate, blood pressure and oxygen saturation), auscultation as well as the measure of cough peak flow.

Discussion: The protocol of this study is the first to evaluate the use of MI-E in hospitalized older adults by the measure of discomfort and relief. In regard to literature on the use of MI-E in patients suffering from neuromuscular pathologies and on the effects of aging on the respiratory system, the hypothesis of the study seems justified. On top of bringing physical benefits to the patient, the study will pave the way for other randomized controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalize in Intensive Care Unit or Pulmonary Unit,
* having airway clearance problem associated with mucus hypersecretion,
* peak expiratory flow (PEF) <280 l/min,
* medical indication for respiratory physical therapy.

Exclusion Criteria:

* contraindication to use of MI-E device (ex. bronchospasm, immediate follow-up to surgery of airway system, chest or abdominal region, untreated pneumothorax, hemodynamic failure, etc.),
* refuse to participate,
* pregnant,
* breastfeeding,
* insufficient cognitive status.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - older adults, inpatients having airway clearance problem associated with mucus hypersecretion and weak or insufficient cough.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Discomfort | The MI-E sessions are realized once in the morning and once in the afternoon on two consecutive days, (4 MI-E sessions totally). Discomfort is evaluated after each MI-E session, (4 evaluations totally).
  Use of a numerical scale of discomfort from 0 to 10, (0 - very comfortable, 10 - extremely uncomfortable). The percentage of sessions being evaluated less than or equal to 6 will be presented.
Relief - change in dyspnea | The MI-E sessions are realized once in the morning and once in the afternoon on two consecutive days, (4 MI-E sessions totally). Relief is evaluated for each session, (4 evaluations totally/8 Borg scores).
  Use of a modified Borg scale to quantify dyspnea, (0 - no dyspnea, 10 - maximal dyspnea). Relief is defined as a change in Borg score of dyspnea before and after each MI-E session.

SECONDARY OUTCOMES:
Heart rate | The MI-E sessions are realized once in the morning and once in the afternoon on two consecutive days, (4 MI-E sessions totally). Heart rate is noted before and after each session, (8 times totally).
  Number of contractions of the heart per minute measured with a standard intensive care unit monitoring devices.
Peak cough flow (PCF) | PCF is measured before and after each session, (8 times totally).
  Measurement of PCF through the peak flow meter.
Respiratory rate | Respiratory rate is noted before and after each session, (8 times totally).
  Number of breaths for one minute measured with a standard intensive care unit monitoring devices.
Blood pressure | Blood pressure is noted before and after each session, (8 times totally).
  Pressure of circulating blood against the walls of blood vessels measured in mmHg with a standard intensive care unit monitoring devices.
Blood oxygen saturation | Blood oxygen saturation is noted before and after each session, (8 times totally).
  Measure of the oxygen level of the blood in percent with a standard intensive care unit monitoring devices.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Estenne, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France